CLINICAL TRIAL: NCT00929916
Title: Efficacy of a Low Volume PEG Purgative (MoviPrep®) Administered Entirely in the Morning Compared to Split Dose (PM/AM) Administration
Brief Title: Comparing Two Different Ways to Take MoviPrep® Before Colonoscopy
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: #08C.251
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Colonoscopy
Keywords: colonoscopy; MoviPrep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AM dosing of MoviPrep®: Take prep morning of exam
- PM/AM dosing of MoviPrep®: half of the volume of prep(1L) solution the evening prior, and half (1L) the morning of, colonoscopy.

SUMMARY:
This study will evaluate whether morning-only dosing of MoviPrep® (2L) for afternoon colonoscopy is as effective as a standard dosing regimen of half of the volume of MoviPrep® (1L) solution the evening prior, and half (1L) the morning of, colonoscopy. MoviPrep® is a low volume (2 liters) polyethylene glycol (PEG)-based purgative that is approved for evening-only or split (evening and morning) dosing to cleanse the colon prior to colonoscopy. Patients undergoing afternoon colonoscopies often have inferior colon cleansing. There is evidence that morning-only purgative administration of large volume PEG (4L) is safe and effective. This study will assess whether administration of a low volume PEG regimen will maintain efficacy and improve tolerance by changing a 2-day preparation procedure into a regimen that is completed in 1 day.

DETAILED DESCRIPTION:
primary objectives

• To compare the efficacy of morning dose only MoviPrep® ("AM Dosing") where one-half of the prep is given 7 hours before colonoscopy and the second half is given 4 hours before colonoscopy, versus split dose (PM/AM) MoviPrep® ("PM/AM Dosing") where one-half of the prep is given at 6pm the night prior to colonoscopy and the second half is given 4 hours before colonoscopy.

Efficacy will be assessed based on cleansing of the entire colon, with successful cleansing defined as a score of excellent or good and unsuccessful cleansing defined as a score of fair or poor.

Secondary objectives

* To assess the tolerability of AM Dosing MoviPrep® versus PM/AM Dosing MoviPrep® based on percentage of prep completed, sleep quality/quantity, future prep choice (same prep or alternative prep described), and incidence and severity (using 11-point Likert scale) of any adverse events (i.e. nausea, vomiting, abdominal pain, bloating, light-headedness).
* To evaluate the safety of each dosing administration based on vitals with orthostatic measures (BP, pulse) on day of colonoscopy.
* To evaluate the effect of colon prep on work and productivity as measured by the degree of interference with work/productivity the day prior to colonoscopy.
* To assess difference between two dosing arms with respect to analysis of right colon cleansing, and overall adenoma detection in terms of number, size, location, histology, and morphology.
* To determine the effect of purgative dosing on procedure efficiency by measuring (a) total procedure time, (b) time from anus to cecum, and (c) withdrawal time (excluding time taken for interventions).
* To evaluate the effect of purgative dosing regimen on amount of flushing required during the procedure (0 = none, 1 = <50 ml, 2 = 50-100 ml, 3 = >100 ml).
* To validate a new grading scale for colon cleansing using the de-identified recordings of colonoscopies performed during this study.

ELIGIBILITY:
Inclusion Criteria:

* Elective out-patients scheduled for afternoon colonoscopy (12 pm or later).

Exclusion Criteria:

* Unable or unwilling to consent
* Age < 18 years
* Pregnant
* Breast feeding
* Gastroparesis - known or suspected
* Chronic nausea or vomiting
* Bowel obstruction
* Hypomotility syndrome: pseudo-obstruction, megacolon, etc.
* Severe constipation (< 1 BM a week)
* Greater than 50% resection of colon
* Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency
* PEG allergy
* Significant psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: out-patients scheduled for afternoon colonoscopy in the Thomas Jefferson GI group
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Comparing the efficacy of AM dose only MoviPrep® (1/2 the prep 7 hrs pre colonoscopy and the second 1/2 4 hrs pre colonoscopy), versus PM/AM where 1/2 of the prep is at 6pm the night prior to colonoscopy and the second half is 4 hours before colonoscopy. | once

SECONDARY OUTCOMES:
To assess the tolerability of AM Dosing MoviPrep® versus PM/AM Dosing MoviPrep® based on % of prep completed, sleep quality/quantity, future prep choice (same prep or alternative prep described), and incidence and severity of any adverse events | once
To evaluate the safety of each dosing administration based on vitals with orthostatic measures (BP, pulse) on day of colonoscopy | once
To evaluate the effect of colon prep on work and productivity as measured by the degree of interference with work/productivity the day prior to colonoscopy. | once
To assess difference between two dosing arms with respect to analysis of right colon cleansing, and overall adenoma detection in terms of number, size, location, histology, and morphology. | once
To determine the effect of purgative dosing on procedure efficiency by measuring (a) total procedure time, (b) time from anus to cecum, and (c) withdrawal time (excluding time taken for interventions). | once
To evaluate the effect of purgative dosing regimen on amount of flushing required during the procedure (0 = none, 1 = <50 ml, 2 = 50-100 ml, 3 = >100 ml). | once
To validate a new grading scale for colon cleansing using the de-identified recordings of colonoscopies performed during this study. | once

CONTACTS AND LOCATIONS:
Overall Officials: David M Kastenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States